CLINICAL TRIAL: NCT02720861
Title: Prevalence of Genetic Polymporphism on RNF213 rs112735431 Gene in Non-cardioemboli Ischemic Cerebrovascular Disease: A Cross-sectional Study in Thai Patients
Brief Title: Prevalence of Genetic Polymporphism on RNF213 rs112735431 Gene in Non-cardioemboli Ischemic Cerebrovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suporn Travanichakul, MD., Neurology Division of Chulalongkorn hospital, Chulalongkorn University
Other Study IDs: COA No.282/2015
Record Dates: First submitted 2016-03-15; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Ischemic Stroke
Keywords: RNF213 rs112735431 Gene; Acute Non-embolic ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non embolic ischemic stroke: acute ischemic stroke from atherosclerosis or lacunar stroke
  Interventions: Genetic: DNA sequencing

INTERVENTIONS:
Genetic: DNA sequencing — withdraw 3m blood from vein only once during the whole design to analyse on DNA sequencing on RNF213 rs112735431 Gene

SUMMARY:
To explore the prevalence of genetic polymorphism on RNF213 rs112735431 gene in non-cardioembolic ischemic cerebrovascular disease in Thai patients.

DETAILED DESCRIPTION:
This is an cross-sectional observational study in Chulalongkorn hospital, to determine the prevalence of genetic polymorphism on RNF213 rs112735431 gene in non-cardioembolic ischemic cerebrovascular disease. Patients who are potentially eligible for study participation will be identified through a chart review of patients who were admitted in Chulalongkorn Hospital for acute ischemic stroke treatment.

ELIGIBILITY:
Inclusion Criteria:

* Nationality in Thailand
* Age equal or more than 18 years
* Clinical and imaging diagnosis of acute ischemic stroke
* Patient consent to participate in the research

Exclusion Criteria:

* High risk for cardioembolic stroke by TOAST classification
* Contraindication for venipuncture
* Pregnancy or breast feeding patient
* History of head and neck radiation
* Down's syndrome
* Marfan syndrome
* Autoimmune disease such as SLE
* Ongoing malignancy or remission of malignancy less than 1year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients of Chulalongkorn hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With RNF213 rs112735431 Gene polymorphism | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suporn Travanichakul, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Suporn Travanichakul, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Not Share